CLINICAL TRIAL: NCT03898648
Title: Behavioral Adaptation to Negative Social Cues in Depressed Patients According to Personal History of Suicide Attempt
Brief Title: Behavioral Adaptation to Negative Social Cues in Depressed Patients According to Personal History of Suicide Attempt- COMPASS
Acronym: COMPASS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the follow up of the last patient has been done
Sponsor: University Hospital, Montpellier (Other)
Collaborators: INSERM U960 - Cognitive Neuroscience Laboratory - Paris, France (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL19_0024
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Depression; History of Suicide Attempt
Keywords: Depression; Suicide attempt; Neuropsychology; Decision- making; Social interaction; Implicit Emotional processing
MeSH Terms: conditions — Depression; Suicide, Attempted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depressed patients with history of suicide attempt (Experimental): Depressed patients with a lifetime history of suicide attempt will be evaluated regarding their behavioral adaptation toward negative social cues.
  Interventions: Other: Waiting room task
- Depressed patients without any history of suicide attempt (Experimental): Depressed patients without history of suicide attempt will be evaluated regarding their behavioral adaptation toward negative social cues.
  Interventions: Other: Waiting room task

INTERVENTIONS:
Other: Waiting room task — The waiting room task consists in a computerized neuropsychological task in which the participant is asked to freely choose a chair to sit in a waiting room. In a row of four chairs, the two in the middle are occupied by two males or females. One of the two subjects sitting either has a neutral face, or express a negative emotion (fear or anger).
  To make their decision, participants must press the "S" keyboard button to go left or the "L" keyboard button to go right in a time limit of 1500 milliseconds.
  One third of the time, the cursor moves in the opposite direction to that requested by the participant. For example, if the subject presses "S", the cursor moves to the right instead of to the left.
  Those reverse trials are used to evaluate their motivation to correct the movement of the cursor.
  The participant will repeat the task 360 times for the assessment to be completed.

SUMMARY:
Social interactions are part of daily life. To decide to interact with someone or not is a routine for humans. To ensure the quality of interpersonal relationships, emotional cues must be taken into account to adapt optimally the investigator's behavior.

Difficulties in interpersonal relationships often trigger suicidal behavior. Suicide attempters are characterized by an impaired decision - making associated with difficulties in familial relationships.

To date, little data on emotional recognition and social decision- making in clinical population is available.

The study aims to compare behavioral response to negative social cues in 82 depressed patients according to their history of suicide attempt using a computerized neuropsychological task.

DETAILED DESCRIPTION:
To identify the nature of the mechanisms involved in social decisions, Mennella and coll. have developed a computerized task (waiting room task) in which the participant is asked to avoid or to approach individuals expressing negative emotional expressions, in this case: anger or fear. In practice, participants have to choose between two chairs to sit in a waiting room in which subjects expressing a neutral face or negative emotions are present. To make this choice they must press a specific keyboard button. In addition to that, in order to evaluate motivation, some of the trials are reversed, meaning that the choice made by the participant will result in the opposite result.

Using this task they have shown that: (1) anger is associated with more avoidance behavior than fear, (2) this behavior is goal- directed and, (3) the higher the level of impulsivity of the subjects, the less able they are to adapt their responses.

The proposed study will use this neuropsychological assessment, the waiting room task, to evaluate if depressed patients would avoid or approach individuals expressing negative facial emotions. The main objective is to compare behavioral adaptation to anger vs neutral cues among depressed patients with and without history of suicide attempt.

The study also aims to :

1. compare behavioral response to fear vs. neutral and anger vs. fear in depressed patients according to suicidal history ;
2. assess the modulation of behavioral adaptation by history of childhood maltreatment, level of impulsivity, anxiodepression and anhedonia;
3. correlate behavioral adaptation to negative cues (anger and fear) with decision-making performances using the Iowa Gambling Task.

The hypothesis is that depressed patients with a history of suicide attempt will exhibit anger specific hyper-responsiveness resulting in an increased avoidance behavior compared to subjects without suicidal history. It is expected that depressed suicide attempters will not have a different emotional reactivity compared to patients without suicidal history for another negative emotion, namely fear.

To that purpose, 82 depressed patients will be recruited in the study. Half of them will have a history of suicide attempt (suicide attempters) while the other half will have none (affective controls). Their participation will consist of an unique visit.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years old
* Meeting the DSM-5 criteria for a current major depressive disorder
* For suicidal patients : having a lifetime history of suicide attempt
* For affective controls : having no personal history of suicide attempt
* Being able to understand the nature, purpose and methodology of the study
* Having signed the informed consent
* Being affiliated to a social security system

Exclusion Criteria:

* Current depressive episode with psychotic characteristics
* Mental retardation or sever medical co-morbidity
* Lifetime Diagnosis of schizophrenia or schizoaffective disorder
* Current manic or hypomanic episode
* Sensory or cognitive disability
* Pregnant or breastfeeding woman
* Deprivation of liberty (by judicial or administrative decision)
* Protection by law (guardianship or curatorship)
* Exclusion period in relation to another protocol
* Inability to understand, speak and write French

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Motivation to avoid anger during the emotional task | At inclusion
  Calculation of the proportion of avoidance vs. approach choices from people expressing anger

SECONDARY OUTCOMES:
Change in the proportion of avoidant choices in reverse trials compared to normal trials | At inclusion
  Computerized calculation of the proportion of avoidance choices in reverse trials and comparison to the proportion calculated in normal trials.
Reaction time before clicking | At inclusion
  Computerized measurement of reaction time before clicking to make the avoidant or approach choice
Reaction time between first and second choices in reverse tests | At inclusion
  Computerized measurement of reaction time between the first choice and the second choice during the reverse condition
Iowa Gambling Test score | At inclusion
  Decision- making impairment assessment with the Iowa Gambling Task. In this task participants are asked to choose between four piles of cards allowing them to earn or lose money. - Among those piles, two are advantageous (little gain and little loss) while the other two are disadvantageous (bigger gain but bigger loss). The goal is to earn as much money as possible. Persistence to choose the disadvantageous piles is interpreted to reflect impulsivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Uhmontpellier, Montpellier, France